CLINICAL TRIAL: NCT04871204
Title: Octreotide Treatment to Improve Nutritional Recovery After Surgery for Patients with Esophageal or Gastric Cancer, a Prospective Randomized Open Label Phase II Study - OTIS
Brief Title: Octreotide Treatment to Improve Nutritional Recovery After Surgery for Patients with Esophageal or Gastric Cancer
Acronym: OTIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fredrik Klevebro (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Sponsor-Investigator, Fredrik Klevebro, Principal Investigator, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OTIS2019_001
Record Dates: First submitted 2021-04-23; First posted 2021-05-04 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: Weight loss; Quality of Life; Nutritional recovery
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Weight Loss | interventions — Octreotide

STUDY DESIGN:
Intervention Model Description: Parallell design with Control arm receiving standard treatment and Experimental arm receiving Octreotide treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Standard treatment
- Octreotide (Experimental): 3 monthly intramuscular injections of 10 mg Octreotide
  Interventions: Drug: Octreotide Injection

INTERVENTIONS:
Drug: Octreotide Injection — 10 mg Sandostatin LAR intramuscular injection
  Arms: Octreotide

SUMMARY:
The aim of the study is to clarify whether octreotide therapy can reduce undesired postoperative weight loss, increase health-related quality of life and improve the appetite after surgery for esophageal or gastric cancer.

DETAILED DESCRIPTION:
Dietary complications are the biggest problem for patients before, during and after surgical treatment. Improved multimodal therapy and centralization of treatment to highly specialized centers have led to an increase in the number of patients surviving with chronic negative effects of esophageal surgery. The scientific state of knowledge about HRQOL and the symptoms of long-term survival of esophageal cancer is limited.

Patient-reported outcome measures (PRUs) are results reported by the patient himself, e.g. HRQOL, remaining symptoms, satisfaction with health care and other problems in daily life. These results have rarely been of importance before but are now increasingly crucial in the evaluation of treatment. It is no longer just about survival for patients with cancer of the esophagus. The aim of the study is to clarify whether octreotide therapy can reduce undesired postoperative weight loss, increase health-related quality of life and improve the appetite after surgery for esophageal or gastric cancer.

Our hypothesis is that intramuscularly administered octreotide can decrease weight loss after gastrectomy or esophagectomy due to cancer and that it may improve postoperative health related quality of life. This study aims to investigate if postoperative eating problems can be reduced by treatment with octreotide in this patient group.

In the first part of the study: Sub study 1, safety, tolerability and feasibility of octreotide treatment will be investigated. Twenty patients diagnosed with esophageal or gastric cancer will receive three monthly injections of 10 mg of Sandostatin LAR depot. Patients will be followed up at 1, 2, 3 and 6 months for monitoring of safety blood parameters, changes in weight, health-related quality of life and adverse events.

In the second part of the study: Sub study 2, efficacy of treatment with octreotide will be studied. 152 patients diagnosed with esophageal or gastric cancer will be randomized 1:1 to post-surgical treatment with octreotide or no treatment. Patients in the active arm will receive three monthly injections of 10 mg of Sandostatin LAR depot. All patients will be followed up at 1, 2, 3 and 6 months in the same manner as in Sub study 1. In this study part gastrointestinal satiety hormones and nutritional evaluation associated quality of life will be studied in addition to body weight, body composition and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologic anatomic analysis (PAD) confirmed esophageal or gastric cancer
2. Gastrectomy or esophagectomy with curative intent
3. ≥18 years of age
4. Signed informed consent
5. Able to comply with the procedures of the study protocol, in the opinion of the investigator
6. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, only after A. leaving a negative result on a highly sensitive pregnancy test, B. are using a highly effective method of contraception during treatment, and C. throughout the study.

Exclusion Criteria:

1. Non-radical operation (defined by macroscopic assessment) or metastatic disease diagnosed at the time of surgery
2. Complications leading to restrictions in postoperative oral intake
3. Advanced comorbidity with ASA score III or more
4. Bradycardia (defined as resting heart rate of under 60 beats per minute)
5. Chronic obstructive pulmonary disease
6. Chronic liver disease
7. Insulinoma
8. Kidney failure
9. Concomitant medication with: cyclosporine, cimetidine, bromocriptine, quinidine, or terfenadine
10. Known or suspected allergy to octreotide
11. Mental inability, reluctance or language difficulties that result in difficulty understanding the meaning of study participation
12. Pregnant or nursing female
13. Participation or recent participation in a clinical study with an investigational product (within the last 3 months). Previous participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Weight change in percent (%) | From baseline before surgery, at 1, 2, 3, and 6 months
  Weight loss in percent (%) from baseline weight before surgery, measured at 1, 2, 3, and 6 months after surgery

SECONDARY OUTCOMES:
Changes in gastrointestinal satiety hormone levels | Baseline, 7 days post-surgery and at 1, 2, 3 and 6 months
  Measurement of S-GLP-1, S-PYY, S-Ghrelin and S-GIP (prior to octreotide administration), measured at baseline, 7 days post-surgery and after 1, 2, 3 and 6 months.
Changes in body composition | Baseline, 1, 2, 3, and 6 months
  Body composition measured in percent (%) body fat (continuously)
Changes in nutritional status - PG-SGA | Baseline, 1, 2, 3, and 6 months
  Nutritional status measured with the questionnaire PG-SGA
Changes in nutritional status - EORTC CAX24 | Baseline, 1, 2, 3, and 6 months
  Nutritional status measured with the questionnaire EORTC CAX24
Health-related Quality of Life - EORTC QLQ-C30 | Baseline, 1, 2, 3 and 6 months
  Health-related Quality of Life (HRQOL) measured using EORTC QLQ-C30 at baseline and at 1, 2, 3 and 6 months after randomization
Health-related Quality of Life - QLQ-OG25 | Baseline, 1, 2, 3 and 6 months
  Health-related Quality of Life (HRQOL) measured using QLQ-OG25 at baseline and at 1, 2, 3 and 6 months after randomization
Percentage (of subjects) in need of enteral nutrition | Baseline, 1, 2, 3 and 6 months
  Percentage (of subjects) in need of enteral nutrition with a jejunostomy feeding catheter or nasogastric tube
Number and type of Adverse Events | From 7 days post-surgery and at 1, 2, 3 and 6 months (continuously)
  Number and type of Adverse Events, including known AEs of Sandostatin LAR depot
Number of patients completing treatment | From first treatment at 7 days post-surgery to last treatment at 2 months
  Number of patients completing treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Klevebro, MD, PhD, Principal Investigator — Center for Upper Gastrointestinal Cancer, Theme Cancer, Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Huddinge, Stockholm, Sweden